CLINICAL TRIAL: NCT03335345
Title: Non-inferiority Study of the Pursuit of Enteral Nutrition Compared to a Strategy of Gastric Emptiness Peri-extubation. Cluster Randomized Trial
Acronym: AMBROISIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHM-2016/S3/07
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Non-inferiority, in Terms of Extubation Failure, Continuation of Enteral Nutrition Before Extubation Versus Gastric Vacuity Peri-extubation
Keywords: Airway Extubation/adverse effects/ Methods; Nutrition; Ventilator Weaning/methods; Intensive care Unit; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maximum gastric void (Other): stopping enteral feeding at least 6 hours before extubation. Suction in the gastric tube (if its size permits) continuously for 6 hours before extubation.
  Interventions: Other: maximum gastric vacuity
- maintaining calorie intake (Other): maintaining enteral caloric intake at the same rate. No aspiration in the gastric tube
  Interventions: Other: maintaining calorie intake

INTERVENTIONS:
Other: maintaining calorie intake — Maintaining enteral caloric intake at the same rate. No aspiration in the gastric tube.
  Arms: maintaining calorie intake
Other: maximum gastric vacuity — stopping enteral feeding at least 6 hours before extubation. Suction in the gastric tube (if its caliber permits) continuously for 6 hours before extubation
  Arms: maximum gastric void

SUMMARY:
Approximately 50 to 60% of ICU patients are subjected to invasive mechanical ventilation-through a tracheal tube. Extubation consists of a key moment for the patient on the road to recovery (1). The extubation failure, is a major disease event. The incidence of extubation failure vary between studies between 10% and 20% of ventilated patients over 48 hours, it is therefore a significant risk including at the individual level. Ultimately, it is observed higher mortality for patients with unsuccessful extubation and this independently of their overall severity (2,3). Among the complications associated with extubation failure observed the occurrence of nosocomial pneumonia. Large-scale epidemiological data, covering nearly half of French ICUs found a risk of nosocomial pneumonia multiplied by a factor of 3 in case of extubation failure. Observing this strong association between nosocomial pneumonia and extubation failure does not presage a causal link. In all cases the onset of pneumonia probably involved in the morbidity and mortality of patients undergoing a failed extubation(4).

Prevention of inhalation may limit congestion and bronchial and lung infection, and thereby reduce the risk of extubation failure. Indeed, the primary pathophysiologic mechanism responsible for nosocomial bronchopulmonary infection is inhalation of oropharyngeal and digestive secretions (5).

This risk of inhalation during intubation motivates the implementation of fasting prior to general anesthesia for elective surgery patients. Indeed, it is recommended to respect a 6-hour fast for solids and 2 hours for liquid (water, fruit juices without pulp, tea or coffee without milk) in this situation (9).

Although the situations are very different from the context of programmed anesthesia and extubation followed by a possible emergency reintubation on failure of extubation in the context of resuscitation, fasting appears as a potential means of limit the inhalation during the period of risk posed extubation and reintubation eventual resuscitation. Nevertheless, it is doubtful of the effectiveness of the single fasting to ensure gastric emptiness during the period of extubation. Indeed, a very large proportion of patients presents the delayed gastric emptying causing prolonged gastric fluid stasis. (10).

Fasting and aspiration of gastric contents through a stomach tube has not, to our knowledge, never been rigorously evaluated in the ICU extubation.

Moreover, the setting of fasting patients is likely to induce significant side effects first and foremost, a charge extra care for paramedics. The other major effect is the calorie deficit induced potential source of infectious complications and a delay in extubation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient in intensive care
* Invasive artificial ventilation for at least 48h at the time of extubation
* Prepyloric enteral feeding for at least 24 hours at the time of extubation
* Age ≥ 18 years

Exclusion Criteria:

* tutorship or curatorship
* Pregnant, parturient or nursing woman
* Patient not affiliated to a social security scheme
* Tracheotomized patient
* Post-pyloric enteral-fed patient (naso-jejunal tube)
* Patient already included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1148 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
reintubation within 7 days after extubation in intensive care. | 7 days

CONTACTS AND LOCATIONS:
Locations (22):
- France (21):
  - Réanimation Médicale-CHU ANGERS, Angers
  - Réanimation médico-chirurgicale-CH BLOIS, Blois
  - Réanimation Chirurgicale-CHU BREST, Brest
  - Réanimation Médicale CHU BREST, Brest
  - Réanimation polyvalente-CH CHARTRES, Chartres
  - Réanimation polyvalente-CH CHOLET, Cholet
  - Réanimation polyvalente-CH DREUX, Dreux
  - Réanimation polyvalente-Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Réanimation médico-chirurgicale- CH LE MANS, Le Mans
  - Réanimation-CH de Pays de MORLAIX, Morlaix
  - Réanimation Chirugicale 2- CHU NANTES, Nantes
  - Réanimation Médicale-CHU NANTES, Nantes
  - Médecine Intensive Réanimation-CH ORLEANS, Orléans
  - Réanimation médico-chirurgicale-CH PARIS ST JOSEPH, Paris
  - Réanimation Médicale-CHU POITIERS, Poitiers
  - Réanimation et Soins Continus-CHI de CORNOUAILLE, Quimper
  - Réanimation Médicale-CHU RENNES, Rennes
  - Réanimation polyvalente-CH SAINT BRIEUC, Saint-Brieuc
  - Réanimation polyvalente-CHG SAINT NAZAIRE, Saint-Nazaire
  - Réanimation Chirurgicale-CHRU TOURS, Tours
  - Réanimation Médicale-CHRU TOURS, Tours
- Réanimation-Brulés-CHU GUADELOUPE, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Landais M, Nay MA, Auchabie J, Hubert N, Frerou A, Yehia A, Mercat A, Jonas M, Martino F, Moriconi M, Courte A, Robert-Edan V, Conia A, Bavozet F, Egreteau PY, Bruel C, Renault A, Huet O, Feller M, Chudeau N, Ferrandiere M, Rebion A, Robert A, Giraudeau B, Reignier J, Thille AW, Tavernier E, Ehrmann S; REVA network and CRICS-TriggerSEP F-CRIN research network. Continued enteral nutrition until extubation compared with fasting before extubation in patients in the intensive care unit: an open-label, cluster-randomised, parallel-group, non-inferiority trial. Lancet Respir Med. 2023 Apr;11(4):319-328. doi: 10.1016/S2213-2600(22)00413-1. Epub 2023 Jan 21. PMID 36693402
- [Derived] Landais M, Nay MA, Auchabie J, Hubert N, Rebion A, Robert A, Giraudeau B, Reignier J, Thille AW, Tavernier E, Ehrmann S. Continuous enteral nutrition compared with a maximal gastric vacuity strategy at the time of extubation in the intensive care unit: protocol for a non-inferiority cluster randomised trial (the Ambroisie Project). BMJ Open. 2021 May 20;11(5):e041799. doi: 10.1136/bmjopen-2020-041799. PMID 34016658